CLINICAL TRIAL: NCT01823484
Title: Effects of AN69 ST Hemofilter on Coagulation During Continuous Renal Replacement Therapy in Critically Ill
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Xiaohua Qiu, physician, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112233
Record Dates: First submitted 2013-03-19; First posted 2013-04-04 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Critically Ill; Acute Kidney Injury; Septic Shock
Keywords: hemofilter; coagulation; CRRT; critically ill
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Shock, Septic; Thrombosis

ARMS (2):
- AN 69 ST hemofilter (Experimental): Use AN 69 ST hemofilter during CRRT
  Interventions: Device: AN 69 ST hemofilter
- AN 69 hemofilter (Active Comparator): Use AN 69 hemofilter during CRRT
  Interventions: Device: AN 69 hemofilter

INTERVENTIONS:
Device: AN 69 ST hemofilter
  Arms: AN 69 ST hemofilter
Device: AN 69 hemofilter
  Arms: AN 69 hemofilter

SUMMARY:
Compared with AN69 hemofilter, AN69 ST hemofilter may prolong the time of hemofilter and decrease the quantity of heparin during continuous renal replacement therapy in critically ill.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years old
* admitted to ICU and need CRRT
* anticipated survival time >72h

Exclusion Criteria:

* allergy to hemofilter or heparin
* heparin associated thrombocytopenia
* pregnancy or lactation
* using other anticoagulate drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The using time of hemofilters | 72h
  The time from the beginning of continuous renal replacement therapy until to the end when continuous renal replacement therapy had to be finished because of clotting or other reasons

SECONDARY OUTCOMES:
activated partial thromboplastin time | every 6h from the begining of continuous renal replacement therapy,up to 72h
  Heparin will be used according to activated partial thromboplastin time, and the quantity will be recorded.

OTHER OUTCOMES:
Number of participants with adverse events during continuous renal replacement therapy | 72h

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaohua Qiu, Nanjing, Jiangsu, China